CLINICAL TRIAL: NCT00580216
Title: A Multicenter, Randomized, Double-blind, Assessor-blind, Non-inferiority Study Comparing the Efficacy and Safety of Once-weekly Subcutaneous Biotinylated Idraparinux (SSR126517E) With Oral Adjusted-dose Warfarin in the Prevention of Stroke and Systemic Thromboembolic Events in Patients With Atrial Fibrillation
Brief Title: Evaluation of Weekly Idrabiotaparinux Sodium Versus Oral Adjusted-dose Warfarin to Prevent Stroke and Systemic Thromboembolic Events in Patients With Atrial Fibrillation
Acronym: BOREALIS-AF
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: early discontinuation based on strategic sponsor decision not driven by any safety concern
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EFC10295; 2007-004817-33 (EudraCT Number)
Record Dates: First submitted 2007-12-21; First posted 2007-12-24 (Estimated); Last update posted 2016-03-21 (Estimated); Status verified 2016-02

CONDITIONS: Atrial Fibrillation
Keywords: stroke; systemic thromboembolic events
MeSH Terms: conditions — Atrial Fibrillation; Stroke | interventions — Warfarin; Avidin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Idrabiotaparinux (Experimental): Idrabiotaparinux sodium, 3.0 mg, once-weekly for 7 weeks followed a maintenance dosing adjusted according to the age and to the renal function for a minimum total treatment duration of 6 months.
  Avidin, 100 mg, at the discretion of the investigator whenever deemed appropriate and possible (ie, life-threatening bleeding, emergency invasive procedure with the potential of uncontrolled bleeding, or overdosage).
  Interventions: Drug: Idrabiotaparinux sodium; Drug: Placebo (for warfarin); Drug: Avidin
- Warfarin (Active Comparator): Warfarin, INR-adjusted dose, for a minimum total treatment duration of 6 months.
  Interventions: Drug: Warfarin; Drug: Placebo (for idrabiotaparinux); Drug: Placebo (for avidin)

INTERVENTIONS:
Drug: Idrabiotaparinux sodium — Pre-filled syringes containing:
  * 0.5 mL for the 3.0 mg dosage;
  * 0.33 mL for the 2.0 mg dosage (maintenance dosage for participants with mild renal impairment and less than 75 years old);
  * 0.25 mL for the 1.5 mg dosage (maintenance dosage for participants with moderate renal impairment or age ≥75 years).
  Subcutaneous injection
  Other Names: SSR126517; Biotinylated idraparinux
  Arms: Idrabiotaparinux
Drug: Warfarin — Capsules with 1 or 5 mg for INR-adjusted dose (INR checked at least once a month)
  Oral administration
  Arms: Warfarin
Drug: Placebo (for idrabiotaparinux) — Matching pre-filled syringes containing:
  * 0.5 mL for the 3.0 mg dosage;
  * 0.33 mL for the 2.0 mg dosage (maintenance dosage for participants with mild renal impairment and less than 75 years old);
  * 0.25 mL for the 1.5 mg dosage (maintenance dosage for participants with moderate renal impairment or age ≥75 years).
  Subcutaneous injection
  Arms: Warfarin
Drug: Placebo (for warfarin) — Warfarin matching capsules
  Oral administration
  Arms: Idrabiotaparinux
Drug: Avidin — Vial containing 105 mg of lyophilized powder for dilution
  Intravenous infusion for 30 minutes
  Other Names: SSR29261
  Arms: Idrabiotaparinux
Drug: Placebo (for avidin) — Vial containing 105 mg of matching lyophilized powder for dissolution
  Intravenous infusion for 30 minutes
  Arms: Warfarin

SUMMARY:
The objective is to evaluate whether once weekly subcutaneous (SC) injection of idrabiotaparinux sodium (biotinylated idraparinux) is at least as efficient to prevent clots in brain and in the other organs than oral international normalized ratio (INR) adjusted-dose warfarin in patients with atrial fibrillation (AF).

DETAILED DESCRIPTION:
The end of the study is defined by a common study end date for all participants, defined as 9 months (39 weeks) after the last participant randomized.

All participants will receive oral warfarin (or matching placebo) and weekly SC injections of idrabiotaparinux sodium (or matching placebo) up to 6 months before the common study end date. All participants are expected to be treated for at least 6 months.

All participants will have then an 6-month observational period after cessation of study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Non valvular atrial fibrillation (AF)
* Indication for long-term Vitamin-K antagonist (VKA) therapy based on the presence of previous ischemic stroke, transient ischemic attack (TIA) or systemic embolism and/or at least two of the following risk factors: hypertension requiring drug treatment, moderately or severely impaired left ventricular function and/or congestive heart failure, age > or = 75 years, diabetes mellitus.

Main exclusion Criteria:

* Indication for VKA other than AF
* Stroke or TIA within previous 5 days
* Transient AF caused by a reversible disorder
* Planned major surgery/trauma or cardioversion within 30 days
* INR > 3 at baseline
* Active bleeding or high risk of bleeding
* Uncontrolled hypertension
* Pregnancy or childbearing potential without proper contraceptive measures or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3773 (Actual)
Dates: Start 2007-12; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Composite of all fatal or non-fatal strokes or non central nervous system (CNS) systemic embolic events (SE) | From randomization up to the end of the treatment period (minimum of 6 months)

SECONDARY OUTCOMES:
Components of the primary study outcome measure: | From randomization up to the end of the treatment period (minimum of 6 months)
Composite of stroke or non CNS SE or myocardial infarction (MI) or venous thromboembolism (VTE) or major bleeding or death | From randomization up to the end of the treatment period (minimum of 6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (538):
- United States (162):
  - Sanofi-Aventis Investigational Site Number 840227, Mobile, Alabama
  - Sanofi-Aventis Investigational Site Number 840209, Tucson, Arizona
  - Sanofi-Aventis Investigational Site Number 840255, Little Rock, Arkansas
  - Sanofi-Aventis Investigational Site Number 840224, Little Rock, Arkansas
  - Sanofi-Aventis Investigational Site Number 840179, Mountain Home, Arkansas
  - Sanofi-Aventis Investigational Site Number 840270, Beverly Hills, California
  - Sanofi-Aventis Investigational Site Number 840278, Beverly Hills, California
  - Sanofi-Aventis Investigational Site Number 840241, Burbank, California
  - Sanofi-Aventis Investigational Site Number 840010, Corona, California
  - Sanofi-Aventis Investigational Site Number 840195, Encino, California
  - Sanofi-Aventis Investigational Site Number 840033, Loma Linda, California
  - Sanofi-Aventis Investigational Site Number 840184, Long Beach, California
  - Sanofi-Aventis Investigational Site Number 840183, Los Banos, California
  - Sanofi-Aventis Investigational Site Number 840272, Northridge, California
  - Sanofi-Aventis Investigational Site Number 840213, Orange, California
  - Sanofi-Aventis Investigational Site Number 840009, Redondo Beach, California
  - Sanofi-Aventis Investigational Site Number 840298, Riverside, California
  - Sanofi-Aventis Investigational Site Number 840264, San Diego, California
  - Sanofi-Aventis Investigational Site Number 840275, San Diego, California
  - Sanofi-Aventis Investigational Site Number 840103, Santa Ana, California
  - Sanofi-Aventis Investigational Site Number 840002, Santa Rosa, California
  - Sanofi-Aventis Investigational Site Number 840111, Torrance, California
  - Sanofi-Aventis Investigational Site Number 840118, Visalia, California
  - Sanofi-Aventis Investigational Site Number 840268, Bridgeport, Connecticut
  - Sanofi-Aventis Investigational Site Number 840246, Bay Pines, Florida
  - Sanofi-Aventis Investigational Site Number 840066, Beach, Florida
  - Sanofi-Aventis Investigational Site Number 840313, Brandon, Florida
  - Sanofi-Aventis Investigational Site Number 840084, Dunnellon, Florida
  - Sanofi-Aventis Investigational Site Number 840138, Fort Lauderdale, Florida
  - Sanofi-Aventis Investigational Site Number 840220, Fort Lauderdale, Florida
  - Sanofi-Aventis Investigational Site Number 840215, Gainesville, Florida
  - Sanofi-Aventis Investigational Site Number 840131, Hollywood, Florida
  - Sanofi-Aventis Investigational Site Number 840161, Hollywood, Florida
  - Sanofi-Aventis Investigational Site Number 840234, Key West, Florida
  - Sanofi-Aventis Investigational Site Number 840112, Lake Mary, Florida
  - Sanofi-Aventis Investigational Site Number 840053, Lakeland, Florida
  - Sanofi-Aventis Investigational Site Number 840198, Melbourne, Florida
  - Sanofi-Aventis Investigational Site Number 840117, Miami, Florida
  - Sanofi-Aventis Investigational Site Number 840003, Niceville, Florida
  - Sanofi-Aventis Investigational Site Number 840230, Ocala, Florida
  - Sanofi-Aventis Investigational Site Number 840202, Orlando, Florida
  - Sanofi-Aventis Investigational Site Number 840306, Orlando, Florida
  - Sanofi-Aventis Investigational Site Number 840022, Ormond Beach, Florida
  - Sanofi-Aventis Investigational Site Number 840110, Palm Harbor, Florida
  - Sanofi-Aventis Investigational Site Number 840211, Plantation, Florida
  - Sanofi-Aventis Investigational Site Number 840116, Sanford, Florida
  - Sanofi-Aventis Investigational Site Number 840243, Spring Hill, Florida
  - Sanofi-Aventis Investigational Site Number 840082, St. Petersburg, Florida
  - Sanofi-Aventis Investigational Site Number 840012, St. Petersburg, Florida
  - Sanofi-Aventis Investigational Site Number 840073, Atlanta, Georgia
  - Sanofi-Aventis Investigational Site Number 840273, Augusta, Georgia
  - Sanofi-Aventis Investigational Site Number 840204, Columbus, Georgia
  - Sanofi-Aventis Investigational Site Number 840290, Columbus, Georgia
  - Sanofi-Aventis Investigational Site Number 840225, Columbus, Georgia
  - Sanofi-Aventis Investigational Site Number 840305, Dunwoody, Georgia
  - Sanofi-Aventis Investigational Site Number 840165, Savannah, Georgia
  - Sanofi-Aventis Investigational Site Number 840130, Idaho Falls, Idaho
  - Sanofi-Aventis Investigational Site Number 840228, Idaho Falls, Idaho
  - Sanofi-Aventis Investigational Site Number 840143, Nampa, Idaho
  - Sanofi-Aventis Investigational Site Number 840221, Chicago, Illinois
  - Sanofi-Aventis Investigational Site Number 840206, Chicago, Illinois
  - Sanofi-Aventis Investigational Site Number 840280, Beaver City, Indiana
  - Sanofi-Aventis Investigational Site Number 840014, Elkhart, Indiana
  - Sanofi-Aventis Investigational Site Number 840249, Wichita, Kansas
  - Sanofi-Aventis Investigational Site Number 840265, Lexington, Kentucky
  - Sanofi-Aventis Investigational Site Number 840047, Alexandria, Louisiana
  - Sanofi-Aventis Investigational Site Number 840218, Jena, Louisiana
  - Sanofi-Aventis Investigational Site Number 840247, Lafayette, Louisiana
  - Sanofi-Aventis Investigational Site Number 840158, Lake Charles, Louisiana
  - Sanofi-Aventis Investigational Site Number 840077, Natchitoches, Louisiana
  - Sanofi-Aventis Investigational Site Number 840259, Shreveport, Louisiana
  - Sanofi-Aventis Investigational Site Number 840231, Shreveport, Louisiana
  - Sanofi-Aventis Investigational Site Number 840232, Shreveport, Louisiana
  - Sanofi-Aventis Investigational Site Number 840145, Auburn, Maine
  - Sanofi-Aventis Investigational Site Number 840017, Baltimore, Maryland
  - Sanofi-Aventis Investigational Site Number 840317, Denton, Maryland
  - Sanofi-Aventis Investigational Site Number 840311, Alpena, Michigan
  - Sanofi-Aventis Investigational Site Number 840276, Brighton, Michigan
  - Sanofi-Aventis Investigational Site Number 840242, Detroit, Michigan
  - Sanofi-Aventis Investigational Site Number 840253, Grand Rapids, Michigan
  - Sanofi-Aventis Investigational Site Number 840137, Saint Clair Shores, Michigan
  - Sanofi-Aventis Investigational Site Number 840134, Saint Cloud, Minnesota
  - Sanofi-Aventis Investigational Site Number 840067, Gulfport, Mississippi
  - Sanofi-Aventis Investigational Site Number 840006, Picayune, Mississippi
  - Sanofi-Aventis Investigational Site Number 840201, St Louis, Missouri
  - Sanofi-Aventis Investigational Site Number 840310, St Louis, Missouri
  - Sanofi-Aventis Investigational Site Number 840200, St Louis, Missouri
  - Sanofi-Aventis Investigational Site Number 840323, St Louis, Missouri
  - Sanofi-Aventis Investigational Site Number 840096, Anaconda, Montana
  - Sanofi-Aventis Investigational Site Number 840008, Butte, Montana
  - Sanofi-Aventis Investigational Site Number 840126, Fremont, Nebraska
  - Sanofi-Aventis Investigational Site Number 840051, Las Vegas, Nevada
  - Sanofi-Aventis Investigational Site Number 840258, Las Vegas, Nevada
  - Sanofi-Aventis Investigational Site Number 840303, Hamilton, New Jersey
  - Sanofi-Aventis Investigational Site Number 840109, Linden, New Jersey
  - Sanofi-Aventis Investigational Site Number 840024, Morristown, New Jersey
  - Sanofi-Aventis Investigational Site Number 840102, Buffalo, New York
  - Sanofi-Aventis Investigational Site Number 840152, Johnson City, New York
  - Sanofi-Aventis Investigational Site Number 840159, Rochester, New York
  - Sanofi-Aventis Investigational Site Number 840284, The Bronx, New York
  - Sanofi-Aventis Investigational Site Number 840056, Westfield, New York
  - Sanofi-Aventis Investigational Site Number 840277, Greensboro, North Carolina
  - Sanofi-Aventis Investigational Site Number 840196, Greensboro, North Carolina
  - Sanofi-Aventis Investigational Site Number 840127, Hickory, North Carolina
  - Sanofi-Aventis Investigational Site Number 840150, Raleigh, North Carolina
  - Sanofi-Aventis Investigational Site Number 840185, Rocky Mount, North Carolina
  - Sanofi-Aventis Investigational Site Number 840020, Fargo, North Dakota
  - Sanofi-Aventis Investigational Site Number 840197, Centerville, Ohio
  - Sanofi-Aventis Investigational Site Number 840074, Cincinnati, Ohio
  - Sanofi-Aventis Investigational Site Number 840146, Cleveland, Ohio
  - Sanofi-Aventis Investigational Site Number 840292, Gallipolis, Ohio
  - Sanofi-Aventis Investigational Site Number 840026, Mason, Ohio
  - Sanofi-Aventis Investigational Site Number 840233, Toledo, Ohio
  - Sanofi-Aventis Investigational Site Number 840064, Wadsworth, Ohio
  - Sanofi-Aventis Investigational Site Number 840045, Oklahoma City, Oklahoma
  - Sanofi-Aventis Investigational Site Number 840133, Tulsa, Oklahoma
  - Sanofi-Aventis Investigational Site Number 840113, Bend, Oregon
  - Sanofi-Aventis Investigational Site Number 840257, Portland, Oregon
  - Sanofi-Aventis Investigational Site Number 840304, Indiana, Pennsylvania
  - Sanofi-Aventis Investigational Site Number 840128, Philadelphia, Pennsylvania
  - Sanofi-Aventis Investigational Site Number 840160, Philadelphia, Pennsylvania
  - Sanofi-Aventis Investigational Site Number 840339, Philadelphia, Pennsylvania
  - Sanofi-Aventis Investigational Site Number 840181, Pittsburgh, Pennsylvania
  - Sanofi-Aventis Investigational Site Number 840229, Scotland, Pennsylvania
  - Sanofi-Aventis Investigational Site Number 840072, Stoneboro, Pennsylvania
  - Sanofi-Aventis Investigational Site Number 840248, Cranston, Rhode Island
  - Sanofi-Aventis Investigational Site Number 840261, Anderson, South Carolina
  - Sanofi-Aventis Investigational Site Number 840297, Anderson, South Carolina
  - Sanofi-Aventis Investigational Site Number 840172, Camden, South Carolina
  - Sanofi-Aventis Investigational Site Number 840168, Columbia, South Carolina
  - Sanofi-Aventis Investigational Site Number 840122, Manning, South Carolina
  - Sanofi-Aventis Investigational Site Number 840085, Newberry, South Carolina
  - Sanofi-Aventis Investigational Site Number 840189, Pelzer, South Carolina
  - Sanofi-Aventis Investigational Site Number 840032, Fort Meade, South Dakota
  - Sanofi-Aventis Investigational Site Number 840062, Athens, Tennessee
  - Sanofi-Aventis Investigational Site Number 840048, Bristol, Tennessee
  - Sanofi-Aventis Investigational Site Number 840052, Bristol, Tennessee
  - Sanofi-Aventis Investigational Site Number 840104, Cleveland, Tennessee
  - Sanofi-Aventis Investigational Site Number 840129, Johnson City, Tennessee
  - Sanofi-Aventis Investigational Site Number 840269, Nashville, Tennessee
  - Sanofi-Aventis Investigational Site Number 840076, Amarillo, Texas
  - Sanofi-Aventis Investigational Site Number 840252, Corsicana, Texas
  - Sanofi-Aventis Investigational Site Number 840286, Houston, Texas
  - Sanofi-Aventis Investigational Site Number 840132, Irving, Texas
  - Sanofi-Aventis Investigational Site Number 840005, Odessa, Texas
  - Sanofi-Aventis Investigational Site Number 840289, Odessa, Texas
  - Sanofi-Aventis Investigational Site Number 840186, San Antonio, Texas
  - Sanofi-Aventis Investigational Site Number 840194, San Antonio, Texas
  - Sanofi-Aventis Investigational Site Number 840236, Temple, Texas
  - Sanofi-Aventis Investigational Site Number 840011, Victoria, Texas
  - Sanofi-Aventis Investigational Site Number 840285, Wichita Falls, Texas
  - Sanofi-Aventis Investigational Site Number 840223, Clinton, Utah
  - Sanofi-Aventis Investigational Site Number 840238, Salt Lake City, Utah
  - Sanofi-Aventis Investigational Site Number 840308, Salt Lake City, Utah
  - Sanofi-Aventis Investigational Site Number 840068, Salem, Virginia
  - Sanofi-Aventis Investigational Site Number 840219, Springfield, Virginia
  - Sanofi-Aventis Investigational Site Number 840058, Everett, Washington
  - Sanofi-Aventis Investigational Site Number 840123, Seattle, Washington
  - Sanofi-Aventis Investigational Site Number 840019, Tacoma, Washington
  - Sanofi-Aventis Investigational Site Number 840256, Beloit, Wisconsin
  - Sanofi-Aventis Investigational Site Number 840293, Madison, Wisconsin
  - Sanofi-Aventis Investigational Site Number 840282, Wauwatosa, Wisconsin
- Argentina (10):
  - Sanofi-Aventis Investigational Site Number 032007, Buenos Aires
  - Sanofi-Aventis Investigational Site Number 032011, Buenos Aires
  - Sanofi-Aventis Investigational Site Number 032001, Buenos Aires
  - Sanofi-Aventis Investigational Site Number 032005, Buenos Aires
  - Sanofi-Aventis Investigational Site Number 032009, Capital Federal
  - Sanofi-Aventis Investigational Site Number 032012, Corrientes
  - Sanofi-Aventis Investigational Site Number 032006, Mar del Plata
  - Sanofi-Aventis Investigational Site Number 032014, Morón
  - Sanofi-Aventis Investigational Site Number 032016, Salta
  - Sanofi-Aventis Investigational Site Number 032010, Zárate
- Australia (8):
  - Sanofi-Aventis Investigational Site Number 036006, Adelaide
  - Sanofi-Aventis Investigational Site Number 036003, Auchenflower
  - Sanofi-Aventis Investigational Site Number 036008, Box Hill
  - Sanofi-Aventis Investigational Site Number 036005, Coffs Harbour
  - Sanofi-Aventis Investigational Site Number 036001, Kippa-Ring
  - Sanofi-Aventis Investigational Site Number 036002, Kippa-Ring
  - Sanofi-Aventis Investigational Site Number 036009, Launceston
  - Sanofi-Aventis Investigational Site Number 036010, Woden
- Austria (2):
  - Sanofi-Aventis Investigational Site Number 040001, Graz
  - Sanofi-Aventis Investigational Site Number 040004, Linz
- Belarus (4):
  - Sanofi-Aventis Investigational Site Number 112001, Minsk
  - Sanofi-Aventis Investigational Site Number 112002, Minsk
  - Sanofi-Aventis Investigational Site Number 112003, Minsk
  - Sanofi-Aventis Investigational Site Number 112005, Minsk
- Brazil (15):
  - Sanofi-Aventis Investigational Site Number 076019, Belo Horizonte
  - Sanofi-Aventis Investigational Site Number 076011, Campina Grande do Sul
  - Sanofi-Aventis Investigational Site Number 076007, Campinas
  - Sanofi-Aventis Investigational Site Number 076013, Campinas
  - Sanofi-Aventis Investigational Site Number 076001, Curitiba
  - Sanofi-Aventis Investigational Site Number 076017, Goiânia
  - Sanofi-Aventis Investigational Site Number 076016, Goiânia
  - Sanofi-Aventis Investigational Site Number 076018, Maceió
  - Sanofi-Aventis Investigational Site Number 076012, Porto Alegre
  - Sanofi-Aventis Investigational Site Number 076008, Porto Alegre
  - Sanofi-Aventis Investigational Site Number 076014, Porto Alegre
  - Sanofi-Aventis Investigational Site Number 076009, Recife
  - Sanofi-Aventis Investigational Site Number 076005, São José do Rio Preto
  - Sanofi-Aventis Investigational Site Number 076010, São Paulo
  - Sanofi-Aventis Investigational Site Number 076015, Uberlândia
- Bulgaria (5):
  - Sanofi-Aventis Investigational Site Number 100004, Pleven
  - Sanofi-Aventis Investigational Site Number 100005, Plovdiv
  - Sanofi-Aventis Investigational Site Number 100001, Sofia
  - Sanofi-Aventis Investigational Site Number 100002, Sofia
  - Sanofi-Aventis Investigational Site Number 100003, Sofia
- Canada (4):
  - Sanofi-Aventis Investigational Site Number 124014, London
  - Sanofi-Aventis Investigational Site Number 124006, Newmarket
  - Sanofi-Aventis Investigational Site Number 124012, Québec
  - Sanofi-Aventis Investigational Site Number 124011, Toronto
- Chile (8):
  - Sanofi-Aventis Investigational Site Number 152007, Santiago
  - Sanofi-Aventis Investigational Site Number 152001, Santiago
  - Sanofi-Aventis Investigational Site Number 152003, Santiago
  - Sanofi-Aventis Investigational Site Number 152004, Santiago
  - Sanofi-Aventis Investigational Site Number 152005, Santiago
  - Sanofi-Aventis Investigational Site Number 152008, Santiago
  - Sanofi-Aventis Investigational Site Number 152009, Viña del Mar
  - Sanofi-Aventis Investigational Site Number 152006, Viña del Mar
- Colombia (5):
  - Sanofi-Aventis Investigational Site Number 170003, Bogotá
  - Sanofi-Aventis Investigational Site Number 170006, Bogotá
  - Sanofi-Aventis Investigational Site Number 170001, Bucaramanga
  - Sanofi-Aventis Investigational Site Number 170005, Envigado-Antioquia
  - Sanofi-Aventis Investigational Site Number 170002, Medellín
- Sanofi-Aventis Investigational Site Number 188004, San José, Costa Rica
- Croatia (3):
  - Sanofi-Aventis Investigational Site Number 191003, Split
  - Sanofi-Aventis Investigational Site Number 191001, Zagreb
  - Sanofi-Aventis Investigational Site Number 191004, Zagreb
- Czechia (10):
  - Sanofi-Aventis Investigational Site Number 203005, Chomutov
  - Sanofi-Aventis Investigational Site Number 203003, Jihlava
  - Sanofi-Aventis Investigational Site Number 203009, Ostrava Vitkovice
  - Sanofi-Aventis Investigational Site Number 203001, Pardubice
  - Sanofi-Aventis Investigational Site Number 203011, Plzen - Bory
  - Sanofi-Aventis Investigational Site Number 203002, Prague
  - Sanofi-Aventis Investigational Site Number 203004, Prague
  - Sanofi-Aventis Investigational Site Number 203010, Prague
  - Sanofi-Aventis Investigational Site Number 203006, Prostějov
  - Sanofi-Aventis Investigational Site Number 203008, Ústí nad Orlicí
- Denmark (7):
  - Sanofi-Aventis Investigational Site Number 208002, Glostrup Municipality
  - Sanofi-Aventis Investigational Site Number 208001, Hellerup
  - Sanofi-Aventis Investigational Site Number 208007, Hvidovre
  - Sanofi-Aventis Investigational Site Number 208003, København S
  - Sanofi-Aventis Investigational Site Number 208004, Odense
  - Sanofi-Aventis Investigational Site Number 208006, Roskilde
  - Sanofi-Aventis Investigational Site Number 208005, Svendborg
- Egypt (4):
  - Sanofi-Aventis Investigational Site Number 818002, Alexandria
  - Sanofi-Aventis Investigational Site Number 818003, Alexandria
  - Sanofi-Aventis Investigational Site Number 818004, Alexandria
  - Sanofi-Aventis Investigational Site Number 818001, Cairo
- Estonia (4):
  - Sanofi-Aventis Investigational Site Number 233003, Tallinn
  - Sanofi-Aventis Investigational Site Number 233004, Tallinn
  - Sanofi-Aventis Investigational Site Number 233001, Tallinn
  - Sanofi-Aventis Investigational Site Number 233002, Tartu
- Sanofi-Aventis Investigational Site Number 246001, Helsinki, Finland
- France (26):
  - Sanofi-Aventis Investigational Site Number 250028, Abbeville
  - Sanofi-Aventis Investigational Site Number 250012, Albi
  - Sanofi-Aventis Investigational Site Number 250034, Allauch
  - Sanofi-Aventis Investigational Site Number 250031, Belfort
  - Sanofi-Aventis Investigational Site Number 250011, Bordeaux
  - Sanofi-Aventis Investigational Site Number 250010, Brest
  - Sanofi-Aventis Investigational Site Number 250021, Brest
  - Sanofi-Aventis Investigational Site Number 250035, Bron
  - Sanofi-Aventis Investigational Site Number 250022, Cholet
  - Sanofi-Aventis Investigational Site Number 250006, Dijon
  - Sanofi-Aventis Investigational Site Number 250018, Dijon
  - Sanofi-Aventis Investigational Site Number 250004, La Rochelle
  - Sanofi-Aventis Investigational Site Number 250029, Le Chesnay
  - Sanofi-Aventis Investigational Site Number 250019, Lille
  - Sanofi-Aventis Investigational Site Number 250015, Lille
  - Sanofi-Aventis Investigational Site Number 250030, Metz-Tessy
  - Sanofi-Aventis Investigational Site Number 250003, Montpellier
  - Sanofi-Aventis Investigational Site Number 250032, Montpellier
  - Sanofi-Aventis Investigational Site Number 250016, Nice
  - Sanofi-Aventis Investigational Site Number 250001, Paris
  - Sanofi-Aventis Investigational Site Number 250014, Paris
  - Sanofi-Aventis Investigational Site Number 250008, Paris
  - Sanofi-Aventis Investigational Site Number 250005, Saint-Etienne
  - Sanofi-Aventis Investigational Site Number 250026, Toulouse
  - Sanofi-Aventis Investigational Site Number 250027, Tours
  - Sanofi-Aventis Investigational Site Number 250002, Vandœuvre-lès-Nancy
- Greece (7):
  - Sanofi-Aventis Investigational Site Number 300009, Athens
  - Sanofi-Aventis Investigational Site Number 300007, Athens
  - Sanofi-Aventis Investigational Site Number 300002, Athens
  - Sanofi-Aventis Investigational Site Number 300005, Athens
  - Sanofi-Aventis Investigational Site Number 300006, Chalcis
  - Sanofi-Aventis Investigational Site Number 300004, Chios
  - Sanofi-Aventis Investigational Site Number 300008, Elefsina
- Guatemala (4):
  - Sanofi-Aventis Investigational Site Number 320002, Guatemala City
  - Sanofi-Aventis Investigational Site Number 320001, Guatemala City
  - Sanofi-Aventis Investigational Site Number 320003, Guatemala City
  - Sanofi-Aventis Investigational Site Number 320004, Guatemala City
- India (17):
  - Sanofi-Aventis Investigational Site Number 356001, Ahmedabad
  - Sanofi-Aventis Investigational Site Number 356010, Ahmedabad
  - Sanofi-Aventis Investigational Site Number 356015, Bangalore
  - Sanofi-Aventis Investigational Site Number 356009, Bangalore
  - Sanofi-Aventis Investigational Site Number 356005, Chennai
  - Sanofi-Aventis Investigational Site Number 356002, Coimbatore
  - Sanofi-Aventis Investigational Site Number 356007, Coimbatore
  - Sanofi-Aventis Investigational Site Number 356013, Lucknow
  - Sanofi-Aventis Investigational Site Number 356006, Lucknow
  - Sanofi-Aventis Investigational Site Number 356017, Mumbai
  - Sanofi-Aventis Investigational Site Number 356014, Mysore
  - Sanofi-Aventis Investigational Site Number 356020, Nashik
  - Sanofi-Aventis Investigational Site Number 356004, New Delhi
  - Sanofi-Aventis Investigational Site Number 356012, New Delhi
  - Sanofi-Aventis Investigational Site Number 356018, Pune
  - Sanofi-Aventis Investigational Site Number 356011, Pune
  - Sanofi-Aventis Investigational Site Number 356003, Secunderabad
- Indonesia (2):
  - Sanofi-Aventis Investigational Site Number 360002, Jakarta
  - Sanofi-Aventis Investigational Site Number 360001, Jakarta
- Israel (10):
  - Sanofi-Aventis Investigational Site Number 376003, Afula
  - Sanofi-Aventis Investigational Site Number 376015, Ashkelon
  - Sanofi-Aventis Investigational Site Number 376001, Giv‘atayim
  - Sanofi-Aventis Investigational Site Number 376007, Haifa
  - Sanofi-Aventis Investigational Site Number 376014, Haifa
  - Sanofi-Aventis Investigational Site Number 376004, Holon
  - Sanofi-Aventis Investigational Site Number 376012, Nahariya
  - Sanofi-Aventis Investigational Site Number 376009, Nazareth
  - Sanofi-Aventis Investigational Site Number 376011, Rehovot
  - Sanofi-Aventis Investigational Site Number 376002, Tel Aviv
- Italy (16):
  - Sanofi-Aventis Investigational Site Number 380015, Ascoli Piceno
  - Sanofi-Aventis Investigational Site Number 380018, Borgo San Lorenzo
  - Sanofi-Aventis Investigational Site Number 380016, Chieti
  - Sanofi-Aventis Investigational Site Number 380005, Fidenza
  - Sanofi-Aventis Investigational Site Number 380010, Merate
  - Sanofi-Aventis Investigational Site Number 380014, Milan
  - Sanofi-Aventis Investigational Site Number 380020, Novara
  - Sanofi-Aventis Investigational Site Number 380001, Padua
  - Sanofi-Aventis Investigational Site Number 380007, Padua
  - Sanofi-Aventis Investigational Site Number 380004, Palermo
  - Sanofi-Aventis Investigational Site Number 380008, Pavia
  - Sanofi-Aventis Investigational Site Number 380021, Perugia
  - Sanofi-Aventis Investigational Site Number 380013, San Daniele del Friuli
  - Sanofi-Aventis Investigational Site Number 380003, Sassari
  - Sanofi-Aventis Investigational Site Number 380011, Torino
  - Sanofi-Aventis Investigational Site Number 380009, Treviso
- Lithuania (4):
  - Sanofi-Aventis Investigational Site Number 440004, Kaunas
  - Sanofi-Aventis Investigational Site Number 440002, Kaunas
  - Sanofi-Aventis Investigational Site Number 440003, Vilnius
  - Sanofi-Aventis Investigational Site Number 440001, Vilnius
- Malaysia (3):
  - Sanofi-Aventis Investigational Site Number 458002, George Town
  - Sanofi-Aventis Investigational Site Number 458001, Kuching
  - Sanofi-Aventis Investigational Site Number 458005, Taiping
- Mexico (10):
  - Sanofi-Aventis Investigational Site Number 484008, Acapulco
  - Sanofi-Aventis Investigational Site Number 484013, Aguascalientes
  - Sanofi-Aventis Investigational Site Number 484016, Aguascalientes
  - Sanofi-Aventis Investigational Site Number 484004, Guadalajara
  - Sanofi-Aventis Investigational Site Number 484007, Guadalajara
  - Sanofi-Aventis Investigational Site Number 484012, Mexico City
  - Sanofi-Aventis Investigational Site Number 484010, Monterrey
  - Sanofi-Aventis Investigational Site Number 484011, San Luis Potosí City
  - Sanofi-Aventis Investigational Site Number 484005, San Luis Potosí City
  - Sanofi-Aventis Investigational Site Number 484003, Veracruz
- Morocco (2):
  - Sanofi-Aventis Investigational Site Number 504001, Marrakesh
  - Sanofi-Aventis Investigational Site Number 504002, Meknes
- Netherlands (25):
  - Sanofi-Aventis Investigational Site Number 528012, Almelo
  - Sanofi-Aventis Investigational Site Number 528030, Amsterdam
  - Sanofi-Aventis Investigational Site Number 528026, Breda
  - Sanofi-Aventis Investigational Site Number 528009, Delft
  - Sanofi-Aventis Investigational Site Number 528027, Ede
  - Sanofi-Aventis Investigational Site Number 528006, Eindhoven
  - Sanofi-Aventis Investigational Site Number 528017, Eindhoven
  - Sanofi-Aventis Investigational Site Number 528016, Gouda
  - Sanofi-Aventis Investigational Site Number 528007, Harderwijk
  - Sanofi-Aventis Investigational Site Number 528001, Heerlen
  - Sanofi-Aventis Investigational Site Number 528024, Heerlen
  - Sanofi-Aventis Investigational Site Number 528003, Hengelo
  - Sanofi-Aventis Investigational Site Number 528010, Hengelo
  - Sanofi-Aventis Investigational Site Number 528031, Hoogeveen
  - Sanofi-Aventis Investigational Site Number 528019, Hoorn
  - Sanofi-Aventis Investigational Site Number 528020, Leeuwarden
  - Sanofi-Aventis Investigational Site Number 528004, Nijmegen
  - Sanofi-Aventis Investigational Site Number 528013, Rotterdam
  - Sanofi-Aventis Investigational Site Number 528022, Sittard-Geleen
  - Sanofi-Aventis Investigational Site Number 528002, Sneek
  - Sanofi-Aventis Investigational Site Number 528035, The Hague
  - Sanofi-Aventis Investigational Site Number 528033, Tilburg
  - Sanofi-Aventis Investigational Site Number 528021, Venlo
  - Sanofi-Aventis Investigational Site Number 528005, Zoetermeer
  - Sanofi-Aventis Investigational Site Number 528025, Zwolle
- New Zealand (3):
  - Sanofi-Aventis Investigational Site Number 554003, Christchurch
  - Sanofi-Aventis Investigational Site Number 554002, Dunedin
  - Sanofi-Aventis Investigational Site Number 554001, Nelson
- Norway (4):
  - Sanofi-Aventis Investigational Site Number 578001, Bergen
  - Sanofi-Aventis Investigational Site Number 578006, Flekkefjord
  - Sanofi-Aventis Investigational Site Number 578005, Lørenskog
  - Sanofi-Aventis Investigational Site Number 578004, Oslo
- Panama (3):
  - Sanofi-Aventis Investigational Site Number 591001, Panama City
  - Sanofi-Aventis Investigational Site Number 591002, Panama City
  - Sanofi-Aventis Investigational Site Number 591003, Panama City
- Peru (5):
  - Sanofi-Aventis Investigational Site Number 604004, Lima
  - Sanofi-Aventis Investigational Site Number 604002, Lima
  - Sanofi-Aventis Investigational Site Number 604001, Lima
  - Sanofi-Aventis Investigational Site Number 604005, Lima
  - Sanofi-Aventis Investigational Site Number 604003, Lima
- Sanofi-Aventis Investigational Site Number 608001, Quezon City, Philippines
- Poland (13):
  - Sanofi-Aventis Investigational Site Number 616013, Chojnice
  - Sanofi-Aventis Investigational Site Number 616011, Gdansk
  - Sanofi-Aventis Investigational Site Number 616014, Gdynia-Redlowo
  - Sanofi-Aventis Investigational Site Number 616009, Katowice
  - Sanofi-Aventis Investigational Site Number 616017, Lodz
  - Sanofi-Aventis Investigational Site Number 616002, Lublin
  - Sanofi-Aventis Investigational Site Number 616012, Ostrowiec Świętokrzyski
  - Sanofi-Aventis Investigational Site Number 616015, Puławy
  - Sanofi-Aventis Investigational Site Number 616007, Torun
  - Sanofi-Aventis Investigational Site Number 616006, Tychy
  - Sanofi-Aventis Investigational Site Number 616001, Warsaw
  - Sanofi-Aventis Investigational Site Number 616010, Warsaw
  - Sanofi-Aventis Investigational Site Number 616008, Wroclaw
- Portugal (4):
  - Sanofi-Aventis Investigational Site Number 620002, Amadora
  - Sanofi-Aventis Investigational Site Number 620007, Braga
  - Sanofi-Aventis Investigational Site Number 620006, Coimbra
  - Sanofi-Aventis Investigational Site Number 620008, Setúbal
- Sanofi-Aventis Investigational Site Number 630001, San Juan, Puerto Rico
- Russia (54):
  - Sanofi-Aventis Investigational Site Number 643033, Barnaul
  - Sanofi-Aventis Investigational Site Number 643040, Chelyabinsk
  - Sanofi-Aventis Investigational Site Number 643050, Chelyabinsk
  - Sanofi-Aventis Investigational Site Number 643036, Chelyabinsk
  - Sanofi-Aventis Investigational Site Number 643009, Kemerovo
  - Sanofi-Aventis Investigational Site Number 643042, Kemerovo
  - Sanofi-Aventis Investigational Site Number 643015, Moscow
  - Sanofi-Aventis Investigational Site Number 643032, Moscow
  - Sanofi-Aventis Investigational Site Number 643007, Moscow
  - Sanofi-Aventis Investigational Site Number 643020, Moscow
  - Sanofi-Aventis Investigational Site Number 643054, Moscow
  - Sanofi-Aventis Investigational Site Number 643052, Moscow
  - Sanofi-Aventis Investigational Site Number 643056, Moscow
  - Sanofi-Aventis Investigational Site Number 643025, Moscow
  - Sanofi-Aventis Investigational Site Number 643053, Moscow
  - Sanofi-Aventis Investigational Site Number 643028, Moscow
  - Sanofi-Aventis Investigational Site Number 643037, Moscow
  - Sanofi-Aventis Investigational Site Number 643001, Moscow
  - Sanofi-Aventis Investigational Site Number 643026, Moscow
  - Sanofi-Aventis Investigational Site Number 643039, Moscow
  - Sanofi-Aventis Investigational Site Number 643011, Moscow
  - Sanofi-Aventis Investigational Site Number 643034, Moscow
  - Sanofi-Aventis Investigational Site Number 643049, Moscow
  - Sanofi-Aventis Investigational Site Number 643030, Moscow
  - Sanofi-Aventis Investigational Site Number 643013, Nizhny Novgorod
  - Sanofi-Aventis Investigational Site Number 643041, Nizniy Novgorod
  - Sanofi-Aventis Investigational Site Number 643051, Novosibirsk
  - Sanofi-Aventis Investigational Site Number 643044, Novosibirsk
  - Sanofi-Aventis Investigational Site Number 643048, Novosibirsk-117
  - Sanofi-Aventis Investigational Site Number 643045, Penza
  - Sanofi-Aventis Investigational Site Number 643023, Perm
  - Sanofi-Aventis Investigational Site Number 643006, Perm
  - Sanofi-Aventis Investigational Site Number 643046, Petrozavodsk
  - Sanofi-Aventis Investigational Site Number 643012, Rostov-on-Don
  - Sanofi-Aventis Investigational Site Number 643008, Ryazan
  - Sanofi-Aventis Investigational Site Number 643022, Saint Petersburg
  - Sanofi-Aventis Investigational Site Number 643038, Saint Petersburg
  - Sanofi-Aventis Investigational Site Number 643016, Saint Petersburg
  - Sanofi-Aventis Investigational Site Number 643017, Saint Petersburg
  - Sanofi-Aventis Investigational Site Number 643047, Saint Petersburg
  - Sanofi-Aventis Investigational Site Number 643018, Saint Petersburg
  - Sanofi-Aventis Investigational Site Number 643010, Saint Petersburg
  - Sanofi-Aventis Investigational Site Number 643027, Saint Petersburg
  - Sanofi-Aventis Investigational Site Number 643002, Saint Petersburg
  - Sanofi-Aventis Investigational Site Number 643029, Samara
  - Sanofi-Aventis Investigational Site Number 643004, Saratov
  - Sanofi-Aventis Investigational Site Number 643005, Saratov
  - Sanofi-Aventis Investigational Site Number 643003, Saratov
  - Sanofi-Aventis Investigational Site Number 643024, Tomsk
  - Sanofi-Aventis Investigational Site Number 643035, Tomsk
  - Sanofi-Aventis Investigational Site Number 643021, Tyumen
  - Sanofi-Aventis Investigational Site Number 643043, Voronezh
  - Sanofi-Aventis Investigational Site Number 643019, Yaroslavl
  - Sanofi-Aventis Investigational Site Number 643031, Yekaterinburg
- Slovakia (5):
  - Sanofi-Aventis Investigational Site Number 703003, Košice
  - Sanofi-Aventis Investigational Site Number 703005, Levice
  - Sanofi-Aventis Investigational Site Number 703004, Nitra
  - Sanofi-Aventis Investigational Site Number 703006, Poprad
  - Sanofi-Aventis Investigational Site Number 703002, Trnava
- South Africa (14):
  - Sanofi-Aventis Investigational Site Number 710011, Bloemfontein
  - Sanofi-Aventis Investigational Site Number 710007, Cape Town
  - Sanofi-Aventis Investigational Site Number 710017, Cape Town
  - Sanofi-Aventis Investigational Site Number 710001, Durban
  - Sanofi-Aventis Investigational Site Number 710012, Durban
  - Sanofi-Aventis Investigational Site Number 710013, eManzimtoti
  - Sanofi-Aventis Investigational Site Number 710009, Johannesburg
  - Sanofi-Aventis Investigational Site Number 710016, Port Elizabeth
  - Sanofi-Aventis Investigational Site Number 710020, Pretoria
  - Sanofi-Aventis Investigational Site Number 710003, Pretoria
  - Sanofi-Aventis Investigational Site Number 710002, Pretoria
  - Sanofi-Aventis Investigational Site Number 710015, Randburg
  - Sanofi-Aventis Investigational Site Number 710014, Scottburgh
  - Sanofi-Aventis Investigational Site Number 710018, Umhlanga
- South Korea (10):
  - Sanofi-Aventis Investigational Site Number 410008, Anyang
  - Sanofi-Aventis Investigational Site Number 410002, Daegu
  - Sanofi-Aventis Investigational Site Number 410006, Goyang
  - Sanofi-Aventis Investigational Site Number 410012, Goyang
  - Sanofi-Aventis Investigational Site Number 410007, Gwangju
  - Sanofi-Aventis Investigational Site Number 410003, Seongnam
  - Sanofi-Aventis Investigational Site Number 410001, Seoul
  - Sanofi-Aventis Investigational Site Number 410004, Seoul
  - Sanofi-Aventis Investigational Site Number 410005, Seoul
  - Sanofi-Aventis Investigational Site Number 410011, Seoul
- Spain (5):
  - Sanofi-Aventis Investigational Site Number 724003, Barcelona
  - Sanofi-Aventis Investigational Site Number 724002, Barcelona
  - Sanofi-Aventis Investigational Site Number 724001, Madrid
  - Sanofi-Aventis Investigational Site Number 724005, Santiago de Compostela
  - Sanofi-Aventis Investigational Site Number 724007, Seville
- Sweden (6):
  - Sanofi-Aventis Investigational Site Number 752003, Gothenburg
  - Sanofi-Aventis Investigational Site Number 752006, Gothenburg
  - Sanofi-Aventis Investigational Site Number 752002, Malmo
  - Sanofi-Aventis Investigational Site Number 752007, Malmo
  - Sanofi-Aventis Investigational Site Number 752004, Östersund
  - Sanofi-Aventis Investigational Site Number 752001, Stockholm
- Taiwan (5):
  - Sanofi-Aventis Investigational Site Number 158003, Kaohsiung City
  - Sanofi-Aventis Investigational Site Number 158002, Taichung
  - Sanofi-Aventis Investigational Site Number 158004, Tainan Hsien
  - Sanofi-Aventis Investigational Site Number 158001, Taipei
  - Sanofi-Aventis Investigational Site Number 158005, Taipei
- Thailand (3):
  - Sanofi-Aventis Investigational Site Number 764001, Bangkok
  - Sanofi-Aventis Investigational Site Number 764002, Bangkok Noi
  - Sanofi-Aventis Investigational Site Number 764003, Muang
- Turkey (Türkiye) (7):
  - Sanofi-Aventis Investigational Site Number 792004, Edirne
  - Sanofi-Aventis Investigational Site Number 792005, Edirne
  - Sanofi-Aventis Investigational Site Number 792002, Istanbul
  - Sanofi-Aventis Investigational Site Number 792001, Istanbul
  - Sanofi-Aventis Investigational Site Number 792003, Istanbul
  - Sanofi-Aventis Investigational Site Number 792006, Kocaeli
  - Sanofi-Aventis Investigational Site Number 792007, Kocaeli
- Ukraine (14):
  - Sanofi-Aventis Investigational Site Number 804013, Dnipro
  - Sanofi-Aventis Investigational Site Number 804015, Dnipro
  - Sanofi-Aventis Investigational Site Number 804005, Dnipropetrovsk
  - Sanofi-Aventis Investigational Site Number 804008, Ivano-Frankivsk
  - Sanofi-Aventis Investigational Site Number 804002, Kharkiv
  - Sanofi-Aventis Investigational Site Number 804004, Kharkiv
  - Sanofi-Aventis Investigational Site Number 804012, Kharkiv
  - Sanofi-Aventis Investigational Site Number 804003, Kiev
  - Sanofi-Aventis Investigational Site Number 804007, Lutsk
  - Sanofi-Aventis Investigational Site Number 804009, Lutsk
  - Sanofi-Aventis Investigational Site Number 804011, Odesa
  - Sanofi-Aventis Investigational Site Number 804010, Ternopil
  - Sanofi-Aventis Investigational Site Number 804006, Uzhhorod
  - Sanofi-Aventis Investigational Site Number 804014, Zaporizhzhia
- Venezuela (2):
  - Sanofi-Aventis Investigational Site Number 862001, Caracas
  - Sanofi-Aventis Investigational Site Number 862002, Maracay

REFERENCES:
- [Result] Buller HR, Halperin J, Hankey GJ, Pillion G, Prins MH, Raskob GE. Comparison of idrabiotaparinux with vitamin K antagonists for prevention of thromboembolism in patients with atrial fibrillation: the Borealis-Atrial Fibrillation Study. J Thromb Haemost. 2014 Jun;12(6):824-30. doi: 10.1111/jth.12546. PMID 24597472